CLINICAL TRIAL: NCT03140631
Title: Use of Protamine for Heparin Reversal After Catheter Ablation of Atrial Fibrillation: A Randomized Trial
Brief Title: Use of Protamine for Heparin Reversal After Catheter Ablation of Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hakan Oral, Director, Cardiac Arrhythmia Service, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00117851
Record Dates: First submitted 2017-04-03; First posted 2017-05-04 (Actual); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation; Catheter Ablation
Keywords: atrial fibrillation; catheter ablation; protamine sulfate; anticoagulation reversal
MeSH Terms: conditions — Atrial Fibrillation | interventions — Protamines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Patients in the control arm will undergo routine post-procedure management prior to removal of vascular sheaths. This includes routine measurements of ACT beginning 90 min after the cessation of the procedure with a goal ACT of <200s or return to pre-procedural baseline prior to sheath removal.
- Protamine (Active Comparator): Patients in the active comparator arm will receive protamine sulfate for rapid reversal of heparin prior to sheath removal. They will first receive a small test dose with close hemodynamic monitoring followed by therapeutic dose if no reaction occurs.ACT levels will then be monitored with a goal ACT of <200s or return to preprocedural baseline prior to removal of vascular sheaths.
  Interventions: Drug: Protamine Sulfate

INTERVENTIONS:
Drug: Protamine Sulfate — Protamine sulfate is a highly basic protein that forms stable compounds with acidic heparin to rapidly neutralize the anticoagulation effects.
  Arms: Protamine

SUMMARY:
The objective of this study is to evaluate the safety, efficacy and efficiency of rapid anticoagulation reversal with protamine sulfate versus routine activated clotting time (ACT) monitoring in patients undergoing catheter based ablation of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patient's referred for radiofrequency ablation (RFA) or cryoablation for atrial fibrillation or atrial flutter (left atrial).
* Age ≥ 18 year
* Patients who are mentally and linguistically able to understand the aim of the trial, comply with the trial protocol, verbally acknowledge the risks, benefits, and alternatives in this trial.

Exclusion Criteria:

* Previous intolerance or allergy to heparin products.
* Current or prior administration of protamine products
* History of femoral access site complications including hematoma, AV fistula, pseudoaneurysm, aneurysm.
* Known lower extremity venous thrombosis.
* Coagulopathy or blood dyscrasias.
* Active malignancy.
* Thrombocytosis (platelet count >600k/ul) or thrombocytopenia (platelet count <100k/ul)
* Planned use of vascular closure device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Oral, MD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 153 patients were enrolled in the trial; however, three patients were removed from the trial before treatment allocation due to physician discretion. These patients never received any treatments and were not included in the analysis.
Groups:
- Control: Patients in the control arm will undergo routine post-procedure management prior to removal of vascular sheaths. This includes routine measurements of activated clotting time (ACT) beginning 90 min after the cessation of the procedure with a goal ACT of <200s or return to pre-procedural baseline prior to sheath removal.
- Protamine: Patients in the active comparator arm will receive protamine sulfate for rapid reversal of heparin prior to sheath removal. They will first receive a small test dose with close hemodynamic monitoring followed by therapeutic dose if no reaction occurs. Activated clotting time (ACT) levels will then be monitored with a goal ACT of <200s or return to preprocedural baseline prior to removal of vascular sheaths.
  Protamine Sulfate: Protamine sulfate is a highly basic protein that forms stable compounds with acidic heparin to rapidly neutralize the anticoagulation effects.
Period: Overall Study
Arm/Group | Control | Protamine
Started | 73 | 77
Completed | 73 | 77
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Protamine: Patients in the active comparator arm will receive protamine sulfate for rapid reversal of heparin prior to sheath removal. They will first receive a small test dose with close hemodynamic monitoring followed by therapeutic dose if no reaction occurs. ACT levels will then be monitored with a goal ACT of <200s or return to preprocedural baseline prior to removal of vascular sheaths.
  Protamine Sulfate: Protamine sulfate is a highly basic protein that forms stable compounds with acidic heparin to rapidly neutralize the anticoagulation effects.
- Total: Total of all reporting groups
Arm/Group | Control | Protamine | Total
Number analyzed (Participants) | 73 | 77 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9) | 63 (12) | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 31 | 56
  Male | 48 | 46 | 94
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kilograms/(meter squared)] | 31 (7) | 32 (6) | 32 (6)
CHAD2Ds2-VASc Score [Mean (Standard Deviation); unit: scores on a scale] — Summation of weighted risk factor points: Congestive Heart Failure (1), Hypertension (1), Age 75 years or older (2), Diabetes Mellitus (1), Stroke/Transient Ischemic Attack/Thromboembolic Event (2), Vascular Disease (1), Age 65 to 74 Years (1), Female Sex (1). The minimum score is 0 and represents the lowest risk of thromboembolic events and 9 is the maximum score and represents the highest risk.
  scores on a scale | 2.2 (1.2) | 2.1 (1.2) | 2.1 (1.2)
Warfarin use [Count of Participants; unit: Participants] — this is a count of the number of participants taking the medication warfarin during study enrollment
  Participants | 14 | 14 | 28
NOAC use [Count of Participants; unit: Participants] — this is a count of the number of participants taking a medication in the class of NOAC (novel oral anticoagulants) at the time of study enrollment
  Participants | 59 | 63 | 122
Hemoglobin [Mean (Standard Deviation); unit: g/dl] | 13.7 (1.6) | 14.4 (1.2) | 14.1 (1.4)
Platelets [Mean (Standard Deviation); unit: 10^3 platelets/mm^3] | 194 (67) | 182 (72) | 188 (70)
INR [Mean (Standard Deviation); unit: ratio] | 1.4 (0.6) | 1.3 (0.5) | 1.4 (0.6)
Creatinine [Mean (Standard Deviation); unit: mg/dl] | 1.0 (0.8) | 1.0 (0.3) | 1.0 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Time to Ambulation
Description: Total length of time from procedural termination to patient ambulation
Time Frame: 0 to 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control | Protamine
Number analyzed (Participants) | 73 | 77
minutes | 480 (92) | 316 (80)
Statistical Analysis 1: Comparison: Control vs Protamine; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Count of Participants Who Experienced Vascular Access Site Complications
Description: Secondary endpoints will include the number of patients who experience a 90-day occurrence of vascular access site complications defined as hematoma formation, aneurysm, pseudoaneurysm, arteriovenous fistula formation, access-site related major bleeding (defined as Bleeding Academic Research Consortium (BARC) type 3a or 5), or procedural intervention for access complications (surgical repair, thrombin injection, et cetera)
Time Frame: checked at 30 and 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Protamine
Number analyzed (Participants) | 73 | 77
Participants
  30 days | 4 | 6
  90 days | 4 | 6
Statistical Analysis 1: Comparison: Control vs Protamine; number of participants who experienced a vascular access site complication at 90 days; Test type: Superiority; p = 0.74, Fisher Exact

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Control | Protamine
All-Cause Mortality (participants affected / at risk) | 1/73 | 0/77
Serious Adverse Events (participants affected / at risk) | 1/73 | 1/77
Other Adverse Events (participants affected / at risk) | 4/73 | 5/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=73) | Protamine (N=77)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Major vascular complication (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=73) | Protamine (N=77)
Minor vascular complication (Vascular disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT03140631/Prot_SAP_000.pdf